CLINICAL TRIAL: NCT06312657
Title: Behavioral Effects of Drugs Inpatient 44: Neurobehavioral Mechanisms of Opioid Choice
Brief Title: Behavioral Effects of Drugs Inpatient 44 Neurobehavioral Mechanisms of Opioid Choice
Acronym: BED(In)(44)
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding ended
Sponsor: Joshua A. Lile, Ph.D. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Joshua A. Lile, Ph.D., Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 81971; R01DA047368 (NIH)
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Money-vs-money task (Experimental)
  Interventions: Behavioral: Drug Cue
- Drug-vs-money task (Experimental)
  Interventions: Behavioral: Money; Drug: Withdrawal

INTERVENTIONS:
Behavioral: Drug Cue — Individualized drug cues paired with choice options reinforced by $0.25
  Arms: Money-vs-money task
Behavioral: Money — Two money values will be tested ($0.25 and $4.00)
  Arms: Drug-vs-money task
Drug: Withdrawal — Participants will be maintained on an opioid agonist. Placebo will be substituted to produce mild-to-moderate withdrawal.
  Arms: Drug-vs-money task

SUMMARY:
The objective of this protocol is to use probabilistic choice tasks, reinforcement learning modeling and fMRI to determine the neurobehavioral mechanisms of decision-making in individuals with opioid use disorder and physical opioid dependence.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must meet criteria for moderate/severe opioid use disorder, report past month opioid misuse, and be physically dependent on short-acting opioids (e.g., heroin, hydromorphone, fentanyl), as evidenced by either urine sample positive for recent opioid use during each visit or if opioid negative, displaying frank withdrawal during screening.
* History of intravenous opioid use.
* Baseline O2 saturation of 95% or greater.
* Between the ages of 18-50 years.
* Female subjects must be using an effective form of birth control (e.g., birth control pills, surgical sterilization, IUD, cervical cap with a spermicide, or abstinence). Urine pregnancy tests will be conducted prior to sessions to ensure that female subjects do not participate if pregnant.
* Able to speak and read English.
* Otherwise healthy.

Exclusion Criteria:

* History of, or current, clinically significant physical disease (e.g., respiratory disease [asthma, COPD, sleep apnea], impaired cardiovascular functioning, seizure disorder or CNS tumors) or current or past history of psychiatric disorder that would limit compliance in the studies, other than substance use disorder.
* Meet diagnostic criteria for psychoactive substance use disorder for substances other than opioids (OUD subjects only) or nicotine/caffeine that would require detoxification (i.e., alcohol, benzodiazepines or barbiturates). Negative urine/breath samples for these substances, and the absence of withdrawal, will be required during screening.
* Contraindications for MRI scanning (e.g., pacemaker, metal implants, claustrophobia, or any other implanted medical device).
* Vision or hearing problems that would preclude completion of experimental tasks.
* Poor venous access.
* Regular use of other medications, with the exception of hormone-based contraceptives for female subjects, daily multivitamins or short-term antibiotic prescriptions.
* At risk for respiratory complications and have predictors of difficult bag mask ventilation (e.g., dentures, very full beard), in case emergency respiratory intervention is needed.
* Seeking treatment for SUD or currently taking buprenorphine or methadone as the primary opioid of use.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Task choices | Tasks will take approximately 45-60 minutes to complete. Participants will complete 5 sessions in which a choice task will be administered.
  Number of choices of each option selected.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-06-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT06312657/ICF_000.pdf